CLINICAL TRIAL: NCT03975010
Title: An Open-label, Randomized, Single-dose, Parallel-group Study to Investigate the PK Profile of Single Dose Buprenorphine Transdermal Patch 20 mg Applied for 3 Days, 40 mg for 3 Days and 40 mg for 4 Days in Chinese Subjects With Chronic Pain
Brief Title: Buprenorphine Transdermal Patches Pharmacokinetic Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BUP14-CN-101
Record Dates: First submitted 2019-05-23; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Naltrexone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BUP TDS 20 mg for 3 days (Experimental): Subjects will be randomized into the arms, use BUP TDS 20 mg for 3 days.
  Interventions: Drug: Buprenorphine Transdermal Patch
- BUP TDS 40 mg for 3 days (Experimental): Subjects will be randomized into the arms, use BUP TDS 40 mg for 3 days.
  Interventions: Drug: Buprenorphine Transdermal Patch
- BUP TDS 40 mg for 4 day (Experimental): Subjects will be randomized into the arms, use BUP TDS 40 mg for 4 days.
  Interventions: Drug: Buprenorphine Transdermal Patch

INTERVENTIONS:
Drug: Buprenorphine Transdermal Patch — This is an open-label, randomised, single-dose, 3 arms study design. Subjects will be randomised into one of 3 arms, in a 1:1:1 ratio, wearing BUP TDS 20 mg for 3 days or 40 mg for 3 days or 40 mg for 4 days. Safety follow-up will be planned at 7~9 days after patch removal.
  The study patch will be applied under the cover of naltrexone to reduce opioid related side-effects. Naltrexone 50 mg will be taken orally every 12 hours, from the evening of Day 00 (13 hours prior to IMP application), until the evening of the patch removal.
  Other Names: Naltrexone Hydrochloride

SUMMARY:
This is an open-label, randomised, single-dose, 3 arms study design.

DETAILED DESCRIPTION:
Subjects will be randomised into one of 3 arms, in a 1:1:1 ratio, wearing BUP TDS 20 mg for 3 days or 40 mg for 3 days or 40 mg for 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female subjects with chronic pain (regardless of the aetiology, cancer-pain excluded), aged 18-55 years (both inclusive).
* The average pain over the last 24 hours should attain ≤ 3 assessed with Numeric Rating Scales (NRS) refer to section 19.5. The pain condition has been lasting for at least 1 month and stable for 7 days prior to entering into the screening and is expected to be stable during the study duration.
* Patients on stable permissible non-opioid analgesics, who in the opinion of the investigator are unlikely to require a change in treatment during the study.
* Karnofsky score of Performance Status ≥ 70.
* Body mass index (BMI) of 19 to 28 kg/m2 (both inclusive); and a total body weight ≥ 50 kg.
* Normal dietary habits (e.g. not vegetarian nor vegan) and willing to only take the food supplied during the period of hospitalization.
* Subjects who are able to read, understand and sign written informed consent prior to study participation and are willing to follow the protocol requirements.
* Female subjects of child bearing potential (less than 1 year post-menopausal) must have a negative urine pregnancy test prior to first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of birth control throughout the study such as sterilisation, implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomised partner. Male subjects (surgical history of bilateral vasectomy excluded) with a partner of child bearing potential must be willing to use adequate and highly effective methods of birth control throughout the study.

Exclusion Criteria:

* Unstable condition of the primary disease of chronic pain, which, in the opinion of the investigator, would complicate the subject's participation in the study (e.g. require initiation of new medication).
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies).
* History of seizures or at risk (i.e. head trauma, epilepsy in family, anamnesis, unclear loss of consciousness).
* Any history of frequent nausea or emesis regardless of aetiology.
* Malignancy or a history of malignancy.
* History of orthostatic hypotension.
* Subjects who have any medical or surgical conditions that might interfere with transdermal absorption, distribution, metabolism, or excretion of drugs.
* Positive results for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibodies (HCV Ab), human immunodeficiency virus antibodies (HIVAb).
* Urine screening before study is positive for opioids, barbiturates, amphetamines, cocaine metabolites, methadone, benzodiazepines, phencyclidine, methamphetamine, or cannabinoids or alcohol breath test is positive.
* Subjects who have a current or past (within 5 years) history of substance or alcohol abuse, or subjects who, in the opinion of the investigator or the sub-investigator, have demonstrated addictive or substance abuse behaviors. Alcohol abuse is defined as regular alcohol consumption exceeding 14 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor).
* Consumption of alcoholic beverages within 48 hours before patch application, and / or refusal to abstain from alcohol throughout the study until at least 48 hours after patch removal.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Use of any medicinal product which inhibits CYP3A4 (e.g. troleandomycin, ketoconazole, gestodene, etc) or induces CYP3A4 (e.g. glucocorticoids, barbiturates, rifampicin,etc) within 4 weeks prior to first patch administration.
* Subjects who are currently taking tricyclic antidepressants or have used tricyclic antidepressants within 4 weeks prior to the first patch administration.
* Subjects taking monoamine oxidase (MAO) inhibiters within the past 14 days prior to the first patch administration
* Subjects taking any opioid drug within the past 14 days prior to the first patch administration.
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days prior to the first patch administration. As an exception, acetaminophen could have been used at doses of ≤1 g/day.
* Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days prior to the screening visit. Concurrent enrolment in another clinical trial is not permitted unless the sole purpose of the other trial is for collection of long-term follow-up/survival data.
* Donated 400 mL or more of blood or blood products within 3 months prior to the start of the study.
* Screening sitting blood pressure (BP) ≥140 mm Hg (systolic) or ≥ 90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is ≥140 mm Hg (systolic) or ≥ 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
* 12-lead ECG demonstrating QTc>450 msec or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS interval exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS interval values should be used to determine the subject's eligibility.
* Subjects who have history of hypersensitivity to opioid analgesic formulations.
* Subjects who have history of hypersensitivity to naltrexone.
* Subjects who have history of hypersensitivity to transdermal delivery system or patch adhesives.
* Subjects with any potential dermatological disorder at a patch application site, e.g. previous and/or current unhealed extensive dermal damage in the area where the patch will be applied (e.g. dermatitis, burns, tattoos, scarring of the skin)
* Subjects who could not discontinue therapy that involved direct heat sources (e.g. heat lamps, electric blankets, heating pads or heated water beds) for the duration of the study
* Subjects with hairy areas who could not, or would not, cut the hair at the patch site for proper placement of the patch
* Special diets such as caffeine or xanthine-containing foods and beverages (including pitaya fruit, mango, grapefruit, coffee, tea, cola, chocolate, grapefruit juice, etc.) should be taken within 48 hours before patch application or during the study.
* Subjects who have difficulty swallowing tablets.
* Subjects who cannot tolerate venipuncture, or subjects who have difficulty in collecting blood, or subjects who have a history of fainting at the sight of blood or needles.
* Unwilling or suspected of not being able to comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic profile of buprenorphine and its primary metabolite, norbuprenorphine_Cmax | from Day0 to Day8 or Day9
  Pharmacokinetic parameters of the prototype buprenorphine, and the primetabolite norbuprenorphine, calculated from plasma concentration-time data following a single application of BUP TDS 20 mg (3 days), 40 mg (3 days) and 40 mg (4 days).
To evaluate the pharmacokinetic profile of buprenorphine and its primary metabolite, norbuprenorphine_AUCt | from Day0 to Day8 or Day9
  Pharmacokinetic parameters of the prototype buprenorphine, and the primetabolite norbuprenorphine, calculated from plasma concentration-time data following a single application of BUP TDS 20 mg (3 days), 40 mg (3 days) and 40 mg (4 days).
To evaluate the pharmacokinetic profile of buprenorphine and its primary metabolite, norbuprenorphine_AUCinf | from Day0 to Day8 or Day9
  Pharmacokinetic parameters of the prototype buprenorphine, and the primetabolite norbuprenorphine, calculated from plasma concentration-time data following a single application of BUP TDS 20 mg (3 days), 40 mg (3 days) and 40 mg (4 days).

CONTACTS AND LOCATIONS:
Overall Officials: Wenping Wang, PhD, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine
Locations (1):
- The Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT03975010/Prot_SAP_000.pdf